CLINICAL TRIAL: NCT00615797
Title: Intravenous Immunoglobulins as Effective Treatment in Sydenham's Chorea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Natal Bioproducts Institute (Unknown)
Responsible Party: Principal Investigator, Jo M Wilmshurst, Prof, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTXO1-2002; REF049/2002
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Sydenham Chorea; Post Streptococcal Movement Disorder
MeSH Terms: conditions — Chorea | interventions — Immunoglobulins, Intravenous; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Group randomized to receive intravenous immunoglobulins in addition to standard therapy for sydenham's chorea
  Interventions: Biological: Intravenous immunoglobulin
- 2 (Placebo Comparator): Group randomized to receive standard intervention for sydenham's chorea alone
  Interventions: Drug: standard interventions penicillin VK and haloperidol

INTERVENTIONS:
Biological: Intravenous immunoglobulin — intravenous immunoglobulin 2g/kg total given over 2 days
  Arms: 1
Drug: standard interventions penicillin VK and haloperidol — Penicillin V K 500mg 12hrly po or 250mg 6 hrly for 10 days IM penicillin to be given at discharge, 1.2 million units if over 30 KG and 600,000 units if weight less than 30 KG haloperidol 0,025mg/kg/day orally in divided doses gradually increasing to a maximum of 0,05mg/kg/day
  Arms: 2

SUMMARY:
Children are at risk of developing an involuntary movement disorder after streptococcal throat infections. Not all children are affected and the severity is individually variable. Affected children have alteration in their behaviour and mood and can become quite compromised in their activities of daily living. The condition is believed to be related to the body having an over efficient immune response to the infection and some of the antibodies made in response to the infection also "attack" centres in the brain controlling movement and mood. Treating these children with immunoglobulins, which "mop up" the antibodies may reverse or improve affected children. This study hopes to clarify this.

DETAILED DESCRIPTION:
INTRODUCTION Acute Rheumatic Fever (ARF), chronic rheumatic heart disease (RHD) and neuropsychiatric/ movement disorders related to group A beta haemolytic streptococcal infections (GABAS) remain major public health problems in South Africa. RHD may require repeated hospital admissions, invasive surgery and often results in premature death. In Africa ARF has a mortality of 2-3%. 1 Likewise, neuropsychiatric disorders such as Sydenham's Chorea (SC) resulting from GABAS result in school difficulties, frequent absenteeism, behaviour problems such as obsessive compulsive disorder and may progress to Tourette Syndrome (personal experience). Patients may suffer from disabling neurologic and psychiatric symptoms many years after their initial episode of ARF (personal experience). The morbidity from these conditions demands enormous resources from the state in terms of medical and surgical treatment and we believe results in preventable stress and suffering to the patient and his or her family. Whilst the ideal goal is primary prevention a measure of secondary prevention has been attained by the use of monthly prophylactic penilente. In cases where ARF has occurred, some further intervention is desirable, to prevent the above complications.

At the Rheumatic Fever Clinic (RFC) at Red Cross Hospital patients with established RHD and old cases of Sydenham's Chorea ( SC) are seen. There are 2-4 new cases of ARF seen per month. ARF remains a notifiable disease but it appears that these new cases are often not notified. (personal communication PAWC health officials) SC is a major manifestation of ARF and following the 1992 update of the modified Jones Criteria, it is sufficient alone to make a diagnosis of ARF.2 The duration of SC ranges from a few weeks to 2 years. Recurrences occur in one third of patients.3 Current treatment of SC is purely symptomatic and whether it resolves in 6 weeks or 2 years is dependent on innate healing mechanisms within the individual. SC is postulated to be mediated through auto- antibodies that mis-recognise neuronal cell components. These complexes then result in an inflammatory response in the basal ganglia with the resultant clinical picture of SC. 3 We hypothesise, that the use of intravenous immunoglobulins ( IVIG) will decrease the number of circulating antibodies thereby decreasing symptom severity and shortening the course of the illness. Prophylactic penicillin must be continued to prevent re-exposure and further formation of antibodies.

AIM We aim to determine whether treatment of SC with IVIG expedites recovery and thus cuts down on morbidity and frequent follow up.

METHOD Our aim is to collect a minimum of 20 patients with acute SC, diagnosed according to the revised Jones Criteria for ARF and with an absence of indicators of other causes of chorea. (Table 1) The study would run for 4 years or until the minimum number are recruited.

Patients would be identified and the chorea would be rated as mild, moderate or severe and all signs of chorea carefully documented as per attached format. (A) Special investigations would be performed (Table 2). Patients with IgA deficiency would be excluded from the study. Informed consent would be obtained. Patients would be randomly selected to receive IVIG and or standard treatment. Each patient will be allocated a code number.

Patients will be admitted to a neurology bed, as usually occurs for the acute management of moderate and severe SC. Patients will be notified.

Standard pharmacological treatment (Table 3) of haloperidol and or sodium valproate will be administered, in addition the trial group will receive IVIG. All patients will commence penicillin prophylaxis. On day two (once the administration of IVIG is complete) the investigator (KW) and a blinded observer (WM) will examine the patient for signs of chorea as per addendum A.

The patient will remain hospitalised until he or she can cope with activities of daily living.

Patients will be reviewed at one month, 3 months, 6 months and 1 year and any other time if necessary, this being consistent with current management. They will be assessed by a blinded observer (WM) and by the chief investigator(KW). Follow up will be at the RFC.

IMI penicillin to be given at discharge, 1.2 million units if over 30 KG and 600,000 units if weight less than 30 KG NB. Improvement of symptoms with IVIG alone, can only be expected after the third week post treatment.5 The aim of this therapy is to shorten the overall course of the illness and to prevent complications.

SAMPLE SIZE We aim to get a minimum of twenty cases, 10 will receive IVIG and 10 standard treatment.

ANALYSIS Aim to get a minimum of 20 new cases. Statistical analysis of the outcome measures will be undertaken.

ETHICS / CONSENT In recent years IVIG have been used successfully and safely in a number of auto-immune conditions. 4 Informed consent will be obtained. Parent consent forms will be available in English, Afrikaans and Xhosa COSTING Salaries. No contract staff or casual assistants would be employed. Already salaried staff would look after the patients. Patients with SC are usually admitted to hospital and all the above treatment is administered except for the administration of IVIG, the assessment of serum gamma-globulins and brain spectroscopy scans (single photon emission computed tomographic scanning). The department of Nuclear Medicine has consented to perform these scans. It has been shown that in hemichorea hypermetabolism occurs in the contralateral basal ganglion and this disappears with resolution of symptoms.8 Nursing duties would remain the same as for current admissions of SC. The only additional nursing duty would be the monitoring of the IV infusion.

The registrars and senior house officers will assist in the management of these patients. As stated earlier ARF is a public health problem in South Africa. It is important therefore that health professionals are aware of the preventative and curative treatments available for the treatment of SC.

ADDENDUM A

ACUTE SYDENHAM'S CHOREA

Patient Details

Present History

Past history

Family and Social History

General examination

Details of CVS

Details of Chorea

To be graded as severe, moderate and mild Severe: unable to ambulate or perform any activity of daily living (ADL) Moderate: ambulate with assistance and able to perform some ADLs Mild: ambulate unaided and able to perform most ADLs Minimal: chorea elicited only during neurological examination (9)

Document whether Hemi-chorea or bilateral

Day 0 = Day of admission Day 1 = treatment commenced

Signs of Chorea Day 0 Day 5 1 mth 3 mth 6 mth 1 year Hypotonia Hungup knee jerks Milkmaid's Grip Darting Tongue Pronator Sign Dishing Spoon hand Hippus Weakness Emotional lability Behaviour disturbances Explosive or indistinct speech Facial Grimaces Generalised restlessness Inappropriate Behaviour eg OCD Shrugging shoulders Writhing TOTAL

(10) Definition of Signs Milkmaid's Grip : inability to maintain contraction when the patient grasps the examiners fingers Darting Tongue: inability to maintain protrusion of the tongue Pronator Sign: tendency to pronate one or both hands when they are extended overhead Dishing Spoon Hand: assumption of a hand posture consisting of wrist flexion, hyperextension of the metacarpophalangeal joints, finger straightening and thumb abduction Hippus: reflex constriction and dilation of pupil Hung up knee jerks: slow to return to pre test position

MEDICATION CHART

Date Medication Dose Side Effects Comments

PATIENT'S STICKER

ELIGIBILITY:
Inclusion Criteria:

* Sydenham chorea moderate to severe (affecting activities of daily living) Raised ASOT titre

Exclusion Criteria:

* Mild Sydenham chorea (not affecting activities of daily living)
* Exclusion of systemic lupus erythematosus
* Exclusion of Wilson's disease
* Exclusion of toxin ingestion

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2002-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
improved scores on the sydenham chorea assessment charts | 6 months

SECONDARY OUTCOMES:
improved quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Walker, MB ChB, Principal Investigator — Red Cross Children's Hospital, University of Cape Town
Locations (1):
- Red Cross Children's Hospital, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Perlmutter SJ, Leitman SF, Garvey MA, Hamburger S, Feldman E, Leonard HL, Swedo SE. Therapeutic plasma exchange and intravenous immunoglobulin for obsessive-compulsive disorder and tic disorders in childhood. Lancet. 1999 Oct 2;354(9185):1153-8. doi: 10.1016/S0140-6736(98)12297-3. PMID 10513708
- [Background] Swedo SE. Sydenham's chorea. A model for childhood autoimmune neuropsychiatric disorders. JAMA. 1994 Dec 14;272(22):1788-91. doi: 10.1001/jama.272.22.1788. No abstract available. PMID 7661914
- [Background] Barron KS, Sher MR, Silverman ED. Intravenous immunoglobulin therapy: magic or black magic. J Rheumatol Suppl. 1992 Apr;33:94-7. PMID 1593608
- [Derived] Gregorowski C, Lochner C, Martin L, Simmons C, Kidd M, Walker K, Wilmshurst JM, Seedat S. Neuropsychological manifestations in children with Sydenham's chorea after adjunct intravenous immunoglobulin and standard treatment. Metab Brain Dis. 2016 Feb;31(1):205-12. doi: 10.1007/s11011-015-9681-1. Epub 2015 May 19. PMID 25987537
- [Derived] Walker K, Brink A, Lawrenson J, Mathiassen W, Wilmshurst JM. Treatment of sydenham chorea with intravenous immunoglobulin. J Child Neurol. 2012 Feb;27(2):147-55. doi: 10.1177/0883073811414058. Epub 2011 Aug 24. PMID 21868369